CLINICAL TRIAL: NCT00107510
Title: Phase II Trial of Docetaxel and Carboplatin Administered Every Two Weeks as Induction Therapy for Stage II or III Breast Cancer
Brief Title: Docetaxel, Carboplatin, and Pegfilgrastim in Treating Patients Who Are Undergoing Surgery for Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0338; NCI-2012-02650 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000420834 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — pegfilgrastim; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + carboplatin + pegfilgrastim + surgery (Experimental): Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Patients also receive pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  No more than 6 weeks after completion of chemotherapy, patients undergo definitive surgery.
  After completion of study therapy, patients are followed every 6 months until disease progression and then annually for up to 5 years. Patients who do not complete all 4 courses of chemotherapy or do not undergo surgery are followed every 6 months for up to 5 years.
  Interventions: Biological: pegfilgrastim; Drug: carboplatin; Drug: docetaxel; Procedure: conventional surgery

INTERVENTIONS:
Biological: pegfilgrastim
Drug: carboplatin
Drug: docetaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving docetaxel and carboplatin together with pegfilgrastim before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving docetaxel and carboplatin together with pegfilgrastim works in treating patients who are undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pathological complete response rate in patients with stage II or III breast cancer treated with neoadjuvant docetaxel, carboplatin, and pegfilgrastim.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the rate of breast-conserving surgery in patients treated with this regimen.
* Determine the clinical response rate in patients treated with this regimen.
* Determine the feasibility of drug administration, in terms of the percent of planned dose actually administered per course, in patients treated with this regimen.
* Determine the proportion of patients with negative pathologic lymph node status after treatment with this regimen.
* Determine the proportion of patients with residual ductal carcinoma in situ after treatment with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Patients also receive pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

No more than 6 weeks after completion of chemotherapy, patients undergo definitive surgery.

After completion of study therapy, patients are followed every 6 months until disease progression and then annually for up to 5 years. Patients who do not complete all 4 courses of chemotherapy or do not undergo surgery are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Clinical stage II or III disease (including T2-4, N0-3)
* No clinical or radiological evidence of distant metastases

  * Isolated supraclavicular lymph node involvement allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * AST or ALT ≤ 5 times upper limit of normal (ULN) AND alkaline phosphatase normal
  * AST or ALT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN
  * AST or ALT normal AND alkaline phosphatase ≤ 5 times ULN

Renal

* Creatinine clearance ≥ 30 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study treatment
* No active unresolved infection
* No history of severe hypersensitivity reaction to docetaxel, carboplatin, or any other drug formulated with polysorbate 80
* No known hypersensitivity to E. coli-derived proteins, filgrastim (G-CSF), or pegfilgrastim
* No peripheral neuropathy ≥ grade 2
* No other invasive malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Surgery

* No prior surgical resection for invasive breast cancer

Other

* No other prior therapy for invasive breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate by histologic evaluation at definitive surgery | Up to 5.5 years

SECONDARY OUTCOMES:
Toxicity profile by CTCAE v3.0 at baseline and each subsequent evaluation | Up to 5.5 years
Rate of breast conserving surgery at definitive surgery after neoadjuvant chemotherapy | Up to 5.5 years
Clinical response rate by clinical examination prior to definitive surgery | Up to 5.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Roy, MD, FACP, Study Chair — Mayo Clinic
Locations (120):
- United States (120):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Background] Reinholz MM, Kitzmann KK, Hillman D, et al.: Differential gene expression in circulating tumor cells between primary and metastatic breast cancer patients. [Abstract] Breast Cancer Res Treat 106 (1): A-5022, S213-4, 2007.
- [Result] Roy V, Pockaj BA, Allred JB, Apsey H, Northfelt DW, Nikcevich D, Mattar B, Perez EA. A Phase II trial of docetaxel and carboplatin administered every 2 weeks as preoperative therapy for stage II or III breast cancer: NCCTG study N0338. Am J Clin Oncol. 2013 Dec;36(6):540-4. doi: 10.1097/COC.0b013e318256f619. PMID 22868240
- [Result] Apsey H, Roy V, Pockaj B, et al.: Surgical practice patterns following NCCTG N0338 "Phase II trial of docetaxel and darboplatin administered every two weeks as induction therapy for stage II and stage III breast cancer". [Abstract] J Clin Oncol 27 (Suppl 15): A-623, 2009.
- [Result] Pockaj BA, Mukherjee P, Tinder TL, et al.: NCCTG N0338: effect of docetaxel and carboplatin on VEGF, PGE2, and immune cells in patients with stage II or III breast cancer. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-5110, 2008.